CLINICAL TRIAL: NCT01887678
Title: Multi-center Double-blind Randomized Controlled Trial to Evaluate Effectiveness and Safety of Co-administered Traumeel® / Zeel® Intra-articular Injections vs Placebo in Patients With Moderate-to-Severe Pain With Osteoarthritis of the Knee
Brief Title: Study of Intra-articular Injections vs Placebo in Patients With Pain From Osteoarthritis of the Knee
Acronym: MOZArT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biologische Heilmittel Heel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C1301
Record Dates: First submitted 2013-06-14; First posted 2013-06-27 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Traumeel S; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traumeel® / Zeel® Injectable Solution (Experimental): Injection volume is 4.2 mL for active study medication (2.0 mL Zeel plus 2.2 mL Traumeel in one intra articular (IA) injection) on treatment days 1, 8 and 15.
  Interventions: Drug: Traumeel® / Zeel® Injectable Solution
- Placebo injectable solution (Placebo Comparator): Injection volume of placebo is 4.2 mL as well (taken from the 10.0 mL vial by unblinded staff member, rest to be kept for drug accountability)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Traumeel® / Zeel® Injectable Solution — Injection volume is 4.2 mL for active study medication (2.0 mL Zeel plus 2.2 mL Traumeel in one IA injection) on treatment days 1, 8 and 15.
  Other Names: Traumeel; Zeel
  Arms: Traumeel® / Zeel® Injectable Solution
Drug: Placebo — Placebo is an injection of Saline
  Other Names: Saline
  Arms: Placebo injectable solution

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of a combined Traumeel® / Zeel® injection against placebo (saline) in patients with moderate-to-severe pain associated with osteoarthritis of the knee.

DETAILED DESCRIPTION:
The primary objective is to demonstrate the superiority of Traumeel® and Zeel® co-administered intra-articular (IA) injections vs placebo IA injections on the change in knee pain in patients with moderate to severe knee pain associated with osteoarthritis.

The secondary objectives are to evaluate reduction of pain and stiffness and change in physical function.

Safety is evaluated by the incidence of treatment emergent adverse events during the treatment period and follow up period for all randomized patients.

ELIGIBILITY:
Inclusion Criteria (Screening Visit 1):

1. Osteoarthritis (OA) of the knee by American College of Rheumatology criteria
2. Men or women between 45-80 years of age.
3. Have documented diagnosis of primary OA of the target knee based on clinical and radiographic criteria (Kellgren-Lawrence Numerical Grading System of Grade 2-3) in the tibial-femoral compartment of the target knee confirmed by standard post-anterior weightbearing X-ray of the knee in full extension taken </= 6 months prior to Visit 1.
4. Currently taking an Nonsteroidal anti-inflammatory drug (NSAID), or acetaminophen on a regular basis (4-7 days/ week) over last 2 weeks prior to Visit 1 and has experienced amelioration of pain on these medications.
5. Must have a 50-foot walk test pain score of less than 40 mm on a 100 mm VAS in the target knee at screening
6. Pain in the non-target (contralateral) knee must not be greater than 30 mm on a 100 mm VAS on 50-foot walk test, and the target knee must be more symptomatic.
7. Willingness to stop all OA treatments.
8. Fully informed of the risks of entering the study and willing to provide written consent to enter the study.
9. Able to understand and be willing to comply with all study requirements, particularly the weekly injection regimen for administration of study drug.
10. Primary complaint is pain immediately following an unassisted 50-foot walk. They must show:

    1. moderate to severe pain score in the target knee as demonstrated by 40 - 90 mm recorded on a 100 mm VAS, and
    2. 20 mm increase in pain from their screening visit pain score (a "flare")
    3. pain in the non-target (contralateral) knee must </= 30 mm on a 100 mm VAS

Exclusion Criteria:

1. Known hypersensitivity or allergy to any of the components of Traumeel or Zeel
2. Known hypersensitivity or allergy to acetaminophen.
3. Has body mass index (BMI) >38 kg/m2.
4. Avoidance of, or aversion to, nonprescription medications.
5. Clinical symptoms of meniscal instability or significant valgus/ varus that requires corrective osteotomy
6. Any major injury or surgery to the target knee in the prior 12 months.
7. One or a combination of the following co-morbidities:

   1. other inflammatory arthropathies, gout or pseudogout within previous 6 months
   2. avascular necrosis
   3. severe bone or joint deformity in target knee
   4. osteonecrosis of either knee
   5. fibromyalgia
   6. pes anserine bursitis
   7. lumbar radiculopathy with referred pain to either knee
   8. neurogenic or vascular claudication
   9. significant anterior knee pain due to diagnosed isolated patella-femoral syndrome in the target knee
   10. target knee joint infection or skin disorder/infection to the area surrounding the knee within previous 6 months
   11. current treatment or treatment of cancer within the previous 2 years (excluding basal cell or squamous cell carcinoma of the skin)
8. Participated in any experimental drug or device study within the prior one (1) month and/or IA injections six (6) months.
9. Referred pain from other joints
10. Significantly debilitating concurrent infection(s)
11. Significant ligamentous instability
12. Any prior viscosupplementation therapy (in target knee) within 6 months prior to Screening
13. Systemic or IA injection of corticosteroids in any joint within 3 months of enrollment
14. Therapy with oral hyaluronic acid products, and/or oral pharmaceutical products containing glucosamine and/or chondroitin sulphate and/or diacerein
15. Therapy with opioids within the last 90 days including intra-dermal delivery systems (patches)
16. Therapy with autologous stem cells
17. Therapy with coumarins such as warfarin, Coumadin; heparin and derivative substances including low molecular weight heparin, synthetic pentasaccharide inhibitors of factor Xa such as fondaparinux and idraparinux; direct factor Xa inhibitors such as rivaroxaban and apixaban; direct thrombin inhibitors such as hirudin, lepirudin, bivalirudin, argatroban and dabigatran.
18. Concomitant inflammatory or other rheumatologic, neurological or cardiovascular diseases which could affect the evaluation of knee pain
19. Ongoing litigation for workers compensation for musculoskeletal injuries or disorders
20. Use of alcohol of more than 4 drinks per day
21. Clinically important axial deviation (varus, valgus) greater than 15 degrees
22. Concomitant severe OA of the hip or other joints, which might interfere with the assessments required by the study
23. Painful knee conditions other than OA (e.g., Paget's disease)
24. Hemiparesis of lower limbs
25. Significant planned surgery to lower limbs, which might interfere with the patient's ability to comply with study requirements
26. Presence of serious gastrointestinal, renal, hepatic, pulmonary, cardiovascular, neurological disease that might interfere with the outcome of the study or the patient's ability to comply with study requirements
27. Presence of infections and/or skin diseases in the area of the injection site such as psoriasis
28. Females who are pregnant or breast-feeding or not using recognized effective contraceptive measures. Females of childbearing potential (including those less than one year post-menopausal) must agree to maintain reliable birth control throughout the study.
29. Clinically significant abnormal laboratory values.
30. Patients who are likely to be non-compliant or uncooperative during the study.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nebojsa Skrepnik, MD, Principal Investigator — Tucson Orthopaedic Institute; Royal Anspach, MD, Principal Investigator — Clinical Research Advantage - Arizona II; Hans Barthel, MD, Principal Investigator — Hans Richard Barthel, M.D., Inc.; Shariar Cohen-Gadol, MD, Principal Investigator — Westlake Medical Research; David Bolshoun, MD, Principal Investigator — Radiant Research Inc. - Denver; Linda Murray, DO, Principal Investigator — Radiant Research Inc; Susan Hole, DO, Principal Investigator — Riverside Clinical Research; Agustin Latorre, MD, Principal Investigator — AppleMed Research, Inc.; Richard Radnovich, DO, Principal Investigator — Injury Care Medical Center; Moges Sisay, MD, Principal Investigator — Global Scientific Innovations; Larkin T Wadsworth, MD, Principal Investigator — Sundance Clinical Research, LLC; Kurian Abraham, MD, Principal Investigator — New Hope Clinical Research; Rakesh Patel, MD, Principal Investigator — PMG Research of Salisbury; George Raad, MD, Principal Investigator — PMG Research of Charlotte; Martin VanCleeff, MD, Principal Investigator — PMG Cary Medical Research; John Rubino, MD, Principal Investigator — PMG Research of Raleigh; Howard R Adelglass, MD, Principal Investigator — Research Across America - NY; Louis Re, MD, Principal Investigator — Manhattan Medical Research; Daniel Whitmer, MD, Principal Investigator — Clinical Inquest Center Ltd.; Jeffrey Klein, MD, Principal Investigator — Radiant Research Inc. - Akron; Rakesh Davit, MD, Principal Investigator — Sterling Research Group, Ltd.; Glenn Smith, DO, Principal Investigator — Hillcrest Clinical Research; Shawn Saylor, DO, Principal Investigator — Blair Orthopedic Associates, Inc; Alex Slandzicki, MD, Principal Investigator — Clinical Research Solutions; Sadia Dar, MD, Principal Investigator — Clinical Research Solutions; Rickey Manning, MD, Principal Investigator — PMG Research of Knoxville; Paul Wakefield, MD, Principal Investigator — PMG Research of Knoxville; Michael R Adams, MD, Principal Investigator — Radiant Research Inc. - Salt Lake City; Teresa Sligh, MD, Principal Investigator — Providence Clinical Research; David. Cardona, MD, Principal Investigator — Universal BioPharma Research Inc.
Locations (29):
- United States (29):
  - Clinical Research Advantage - Arizona II, Phoenix, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Universal BioPharma Research Inc., Dinuba, California
  - Providence Clinical Research, North Hollywood, California
  - Hans Richard Barthel, M.D., Inc., Santa Barbara, California
  - Westlake Medical Research, Westlake Village, California
  - Radiant Research Inc. - Denver, Denver, Colorado
  - Riverside Clinical Research, Edgewater, Florida
  - AppleMed Research, Inc., Miami, Florida
  - Radiant Research Inc., Pinellas Park, Florida
  - Injury Care Medical Center, Boise, Idaho
  - Global Scientific Innovations, Evansville, Indiana
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Manhattan Medical Research, New York, New York
  - Research Across America - NY, New York, New York
  - PMG Cary Medical Research, Cary, North Carolina
  - New Hope Clinical Research, Charlotte, North Carolina
  - PMG Research of Charlotte, Charlotte, North Carolina
  - PMG Research of Raleigh, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Radiant Research Inc. - Akron, Akron, Ohio
  - Sterling Research Group, Ltd, Cincinnati, Ohio
  - Clinical Inquest Center Ltd., Dayton, Ohio
  - Hillcrest Clinical Research, Oklahoma City, Oklahoma
  - Blair Orthopedic Associates, Inc., Altoona, Pennsylvania
  - Clinical Research Solutions, Franklin, Tennessee
  - PMG Research of Knoxville, Knoxville, Tennessee
  - Clinical Research Solutions, Smyrna, Tennessee
  - Radiant Research Inc. - Salt Lake City, Salt Lake City, Utah

REFERENCES:
- [Result] Lozada CJ, del Rio E, Reitberg DP, Smith RA, Kahn CB, Moskowitz RW. A double-blind, randomized, saline-controlled study of the efficacy and safety of co-administered intra-articular injections of Tr14 and Ze14 for treatment of painful osteoarthritis of the knee: The MOZArT trial. Eur J Integr Med 2017;13:54-63. DOI: 10.1016/j.eujim.2017.07.005;

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 28 investigational sites in the United States (US) entered at least one patient into the study database, 24 sites randomized at least one patient, 4 sites had Lead-In screening failures only.
Pre-assignment Details: In total, 287 patients were enrolled into the study, 55 of them were Lead-In screening failures and therefore were not included.
Groups:
- Co-administered Traumeel® and Zeel®: Patients with documented diagnosis of primary osteoarthritis of the based on clinical and radiographic criteria (Kellgren-Lawrence Numerical Grading System of Grade 2-3) in the tibial-femoral compartment with an age of between 45 to 80 years and the ability to understand the explanations and instructions given by the study physician got a Traumeel/Zeel injection solution administered once weekly into the target knee on Study Days 1, 8 and 15.
- Placebo Injectable Solution: Patients with documented diagnosis of primary osteoarthritis of the based on clinical and radiographic criteria (Kellgren-Lawrence Numerical Grading System of Grade 2-3) in the tibial-femoral compartment with an age of between 45 to 80 years and the ability to understand the explanations and instructions given by the study physician got a placebo injection solution administered once weekly into the target knee on Study Days 1, 8 and 15.
Period: Overall Study
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Started | 119 | 113
Completed | 102 | 85
Not Completed | 17 | 28
Not completed — Adverse Event | 4 | 6
Not completed — Exceeded rescue medication dosage | 4 | 5
Not completed — Withdrawal of consent | 3 | 4
Not completed — Lost to Follow-up | 4 | 2
Not completed — Deterioration of clinical condition | 0 | 4
Not completed — Lack of Efficacy | 1 | 2
Not completed — Non-compliance | 0 | 3
Not completed — Specified | 1 | 2

BASELINE CHARACTERISTICS:
Population: In total, 287 patients were enrolled into the study, 55 of them were Lead-In screening failures; therefore, 232 patients could be randomized. 119 patients were randomized to Traumeel/Zeel and 113 patients to Placebo and all randomized patients were included in the Safety Set.
Groups:
- Placebo Injectable Solution: At baseline, patients with documented diagnosis of primary osteoarthritis of the based on clinical and radiographic criteria (Kellgren-Lawrence Numerical Grading System of Grade 2-3) in the tibial-femoral compartment with an age of between 45 to 80 years and the ability to understand the explanations and instructions given by the study physician got a placebo injection solution administered once weekly into the target knee on Study Days 1, 8 and 15.
- Total: Total of all reporting groups
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution | Total
Number analyzed (Participants) | 119 | 113 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.11) | 59.7 (8.68) | 60.2 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 46 | 89
  Male | 76 | 67 | 143
Region of Enrollment [Number; unit: participants]
  United States | 119 | 113 | 232

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Pain as Measured by the WOMAC Osteoarthritis (OA) Index Pain Subscale (Section A, Items #1-5) Measured by 100 mm VAS
Description: Changes of the target (treated) knee were assessed using the Western Ontario and McMaster Universities Osteoarthritis Index version 3.1 (WOMAC OA) whereby patients self-assessed 24 parameters on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) where 0 corresponded to 'None' and 100 to 'Extreme'. To assess pain, scores from WOMAC Section A, items 1 to 5 are averaged to yield the Pain Subscale total score. At Study Days 1, 8 and 15 where injections were administered, this was to be done before injection. A two-sided test of equality of the study drug (Traumeel®-Zeel®) and Placebo at level 0.05 was computed using an analysis of covariance (ANCOVA) model with treatment group as qualitative factor and the corresponding Baseline value of the primary efficacy variable as a covariate. The test decision was based on the (two-sided) p-value for the corresponding test of no treatment difference.
Time Frame: from Baseline (Day 1, predose) to End of Study Visit (up to Day 119)
Population: 119 patients were randomized to Traumeel/Zeel and 113 to Placebo and all were included in the Safety Set. Two patients in each group could not be evaluated for primary efficacy. 117 patients in Traumeel/Zeel and 111 patients in Placebo formed the Full Analysis - efficacy. For missing values, Last-observation carried forward (LOCF) was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
units on a scale | -32.0 (26.88) | -25.5 (24.08)
Statistical Analysis 1: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Test type: Superiority or Other; p = 0.0383, ANCOVA; Least Square = -6.37, 95% CI 2-sided [-12.40 to -0.35], Standard Error of Mean 3.06 — A negative value of the Least Square mean difference indicates a result in favor of Traumeel-Zeel

2. Secondary Outcome: Pain Subscore (WOMAC Section A, Items #1-5) Measured by 100 mm VAS
Description: Changes of the target (treated) knee were assessed using the Western Ontario and McMaster Universities Osteoarthritis Index version 3.1 (WOMAC OA) whereby patients self-assessed 24 parameters on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) where 0 corresponded to 'None' and 100 to 'Extreme'. To assess pain, scores from WOMAC Section A, items 1 to 5 are averaged to yield the Pain Subscale total score. At Study Days 1, 8 and 15 where injections were administered, this was to be done before injection. Changes in pain subscore were analyzed by using an analysis of covariance (ANCOVA) model with treatment group as qualitative factor and Baseline value as a covariate.
Time Frame: from Baseline to post-Baseline visits except End of Study Visit (up to day 105)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
units on a scale
  Day 8±1 | -15.8 (18.65) | -13.6 (19.11)
  Day 15±1 | -24.4 (24.31) | -18.5 (20.02)
  Day 43±3 | -26.8 (26.12) | -21.5 (21.62)
  Day 29±3 | -29.7 (26.65) | -22.4 (22.33)
  Day 57±3 | -30.4 (26.69) | -22.7 (23.37)
  Day 71±3 | -31.0 (26.23) | -23.3 (24.38)
  Day 85±3 | -31.1 (26.63) | 24.7 (24.57)
Statistical Analysis 1: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 8±1; Test type: Superiority or Other; p = 0.3715, ANCOVA; Least Squares = -2.15, 95% CI 2-sided [-6.89 to 2.58]
Statistical Analysis 2: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 15±1; Test type: Superiority or Other; p = 0.0293, ANCOVA; Least Square = -5.87, 95% CI 2-sided [-11.15 to -0.60]
Statistical Analysis 3: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 29±3; Test type: Superiority or Other; p = 0.0686, ANCOVA; Least Squares = -5.24, 95% CI 2-sided [-10.88 to 0.40]
Statistical Analysis 4: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 43±3; Test type: Superiority or Other; p = 0.0150, ANCOVA; Least Squares = -7.25, 95% CI 2-sided [-13.08 to -1.42]
Statistical Analysis 5: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 57±3; Test type: Superiority or Other; p = 0.0134, ANCOVA; Least Squares = -7.56, 95% CI 2-sided [-13.54 to -1.58]
Statistical Analysis 6: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 71±3; Test type: Superiority or Other; p = 0.0121, Least Squares; Least Squares = -7.60, 95% CI 2-sided [-13.52 to -1.68]
Statistical Analysis 7: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 85±3; Test type: Superiority or Other; p = 0.0376, ANCOVA; Least Squares = -6.32, 95% CI 2-sided [-12.28 to -0.37]

3. Secondary Outcome: Stiffness Subscore (WOMAC Section B, Items #6-7) Measured by 100 mm VAS
Description: Changes of the target (treated) knee were assessed using the Western Ontario and McMaster Universities Osteoarthritis Index version 3.1 (WOMAC OA) whereby patients self-assessed parameters on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) where 0 corresponded to 'None' and 100 to 'Extreme'. To assess stiffness, scores from WOMAC Section B, items 6 to 7 are averaged to yield the Stiffness Subscale total score. At Study Days 1, 8 and 15 where injections were administered, this was to be done before injection. Changes in stiffness score were analyzed by using an analysis of covariance (ANCOVA) model with treatment group as qualitative factor and Baseline value as a covariate.
Time Frame: from Baseline (Day 1, predose) to End of Study Visit (up to Day 119)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
units on a scale | -34.1 (28.16) | -28.2 (25.73)
Statistical Analysis 1: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Test type: Superiority or Other; p = 0.1373, ANCOVA; Least Squares = -4.76, 95% CI 2-sided [-11.05 to 1.53]

4. Secondary Outcome: Physical Function Bubscore (WOMAC Section C, Items #8-24) Recorded on 100 mm VAS
Description: Changes of the target (treated) knee were assessed using the Western Ontario and McMaster Universities Osteoarthritis Index version 3.1 (WOMAC OA) whereby patients self-assessed 24 parameters on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) where 0 corresponded to 'None' and 100 to 'Extreme'. To assess physical function, scores from WOMAC Section C, items 8 to 24 are averaged to yield the Physical Function Subscale total score. At Study Days 1, 8 and 15 where injections were administered, this was to be done before injection. Changes in Physical Function subscore were analyzed by using an analysis of covariance (ANCOVA) model with treatment group as qualitative factor and Baseline value as a covariate.
Time Frame: from Baseline (Day 1, predose) to End of Study Visit (up to Day 119)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 110
units on a scale | -31.1 (27.38) | -26.9 (24.40)
Statistical Analysis 1: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Test type: Superiority or Other; p = 0.1715, ANCOVA; Least Squares = -4.24, 95% CI 2-sided [-10.33 to 1.85]

5. Secondary Outcome: Total WOMAC Score (All Subscales) Recorded on 100 mm VAS
Description: Changes of the target (treated) knee were assessed using the Western Ontario and McMaster Universities Osteoarthritis Index version 3.1 (WOMAC OA) whereby patients self-assessed 24 parameters on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) where 0 corresponded to 'None' and 100 to 'Extreme'. A total WOMAC score was computed by averaging all 24 possible responses. At Study Days 1, 8 and 15 where injections were administered, this was to be done before injection. Changes in total WOMAC score were analyzed by using an analysis of covariance (ANCOVA) model with treatment group as qualitative factor and Baseline value as a covariate.
Time Frame: from Baseline (Day 1, predose) to End of Study Visit (up to Day 119)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 110
units on a scale | -31.5 (26.94) | -26.7 (24.14)
Statistical Analysis 1: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Test type: Superiority or Other; p = 0.1211, ANCOVA; Least Squares = -4.77, 95% CI 2-sided [-10.82 to 1.27]

6. Secondary Outcome: Patient Global Assessment (PGA)
Description: Patients made an overall Global Assessment of the knee osteoarthritis with the assessment stages "Very good", "Good", "Fair", "Poor" and "Very poor".
Time Frame: from Baseline (Day 1, predose)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
participants
  Very Good | 1 | 0
  Good | 6 | 7
  Fair | 62 | 59
  Poor | 39 | 43
  Very Poor | 8 | 2
  Missing | 1 | 0

7. Secondary Outcome: Patient Global Assessment (PGA)
Description: as for outcome 6
Time Frame: End of Study Visit (up to Day 119)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
participants
  Very Good | 30 | 22
  Good | 49 | 39
  Fair | 31 | 38
  Poor | 6 | 11
  Very Poor | 1 | 1
  Missing | 0 | 0

8. Secondary Outcome: Physician Global Assessment (PhGA)
Description: Study Physicians made an overall Global Assessment of the knee osteoarthritis with the assessment stages "Very good", "Good", "Fair", "Poor" and "Very poor".
Time Frame: Baseline (Day 1, predose)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
participants
  Very Good | 0 | 0
  Good | 7 | 7
  Fair | 73 | 77
  Poor | 34 | 27
  Very Poor | 3 | 0
  Missing | 0 | 0

9. Secondary Outcome: Physician Global Assessment (PhGA)
Description: as for outcome 8
Time Frame: End of Study Visit (up to Day 119)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
participants
  Very Good | 28 | 20
  Good | 51 | 38
  Fair | 34 | 47
  Poor | 4 | 4
  Very Poor | 0 | 2
  Missing | 0 | 0

10. Secondary Outcome: Pain Immediately Following the 50-foot Walk (100 mm VAS)
Description: Changes of the target (treated) knee pain following a 50 feet walk self-assessed by the patients on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) where 0 corresponded to 'None' and 100 to 'Extreme'.
Time Frame: Baseline (Day 1, predose) to post-Baseline visits (up to day 119)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
units on a scale
  Day 8±1 | -26.5 (22.39) | -21.1 (22.09)
  Day 15±1 | -37.4 (23.80) | -26.5 (21.97)
  Day 29±3 | -38.1 (25.37) | -30.7 (24.14)
  Day 43±3 | -42.3 (25.13) | -32.9 (24.45)
  Day 57±3 | -43.0 (25.04) | -33.6 (25.32)
  Day 71±3 | -42.6 (25.31) | -35.1 (23.69)
  Day 85±3 | -41.3 (27.29) | -35.0 (24.38)
  Day 119±3 | -42.3 (26.33) | -36.7 (24.53)
Statistical Analysis 1: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 8±1; Test type: Superiority or Other; p = 0.1128, ANCOVA; Least Squares = -4.97, 95% CI 2-sided [-11.12 to 1.18]
Statistical Analysis 2: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 15±1; Test type: Superiority or Other; p = 0.0013, ANCOVA; Least Squares = -10.49, 95% CI 2-sided [-16.85 to -4.13]
Statistical Analysis 3: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 29±3; Test type: Superiority or Other; p = 0.0472, ANCOVA; Least Squares = -6.89, 95% CI 2-sided [-13.69 to -0.09]
Statistical Analysis 4: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 43±3; Test type: Superiority or Other; p = 0.0109, ANCOVA; Least Squares = -8.82, 95% CI 2-sided [-15.60 to -2.05]
Statistical Analysis 5: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 57±3; Test type: Superiority or Other; p = 0.0123, ANCOVA; Least Squares = -8.88, 95% CI 2-sided [-15.80 to -1.95]
Statistical Analysis 6: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 71±3; Test type: Superiority or Other; p = 0.0425, ANCOVA; Least Squares = -6.88, 95% CI 2-sided [-13.52 to -0.23]
Statistical Analysis 7: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 85±3; Test type: Superiority or Other; p = 0.1199, ANCOVA; Least Squares = -5.51, 95% CI 2-sided [-12.47 to 1.45]
Statistical Analysis 8: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 119±3; Test type: Superiority or Other; p = 0.1575, ANCOVA; Least Squares = -4.96, 95% CI 2-sided [-11.86 to 1.93]

11. Secondary Outcome: Time to Walking (50-foot Walk Test)
Description: Changes in time to walk 50 feet (seconds)
Time Frame: Baseline (Day 1, predose) to post-Baseline visits (up to day 119)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
seconds
  Day 8±1 | -2.8 (7.38) | -2.5 (5.91)
  Day 15±1 | -3.0 (7.25) | -2.7 (6.90)
  Day 29±3 | -3.7 (8.28) | -3.5 (7.94)
  Day 43±3 | -4.4 (9.23) | -3.9 (8.05)
  Day 57±3 | -4.1 (8.24) | -3.7 (9.02)
  Day 71±3 | -4.6 (9.59) | -4.3 (9.63)
  Day 85±3 | -4.6 (9.84) | -4.9 (10.26)
  Day 119±3 | -4.8 (9.66) | -4.6 (10.24)
Statistical Analysis 1: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 8±1; Test type: Superiority or Other; p = 0.6346, ANCOVA; Least Squares = -0.28, 95% CI 2-sided [-1.45 to 0.89]
Statistical Analysis 2: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 15±1; Test type: Superiority or Other; p = 0.6458, ANCOVA; Least Squares = -0.28, 95% CI 2-sided [-1.49 to 0.92]
Statistical Analysis 3: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 29±3; Test type: Superiority or Other; p = 0.7581, ANCOVA; Least Squares = -0.18, 95% CI 2-sided [-1.35 to 0.99]
Statistical Analysis 4: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 43±3; Test type: Superiority or Other; p = 0.3350, ANCOVA; Least Squares = -0.49, 95% CI 2-sided [-1.48 to 0.51]
Statistical Analysis 5: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 57±3; Test type: Superiority or Other; p = 0.4419, ANCOVA; Least Squares = -0.40, 95% CI 2-sided [-1.44 to 0.63]
Statistical Analysis 6: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 71±3; Test type: Superiority or Other; p = 0.4460, ANCOVA; Least Squares = -0.37, 95% CI 2-sided [-1.32 to 0.58]
Statistical Analysis 7: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 85±3; Test type: Superiority or Other; p = 0.6552, ANCOVA; Least Squares = 0.25, 95% CI 2-sided [-0.84 to 1.33]
Statistical Analysis 8: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; Day 119±3; Test type: Superiority or Other; p = 0.7443, ANCOVA; Least Squares = -0.19, 95% CI 2-sided [-1.33 to 0.95]

12. Other Pre Specified Outcome: Serious Adverse Events
Description: Total number of patients affected.
Time Frame: Start of Lead-In period until individual study end, up to 16 weeks.
Population: 119 patients were randomized to Traumeel/Zeel and 113 patients to Placebo and all randomized patients were included in the Safety Set. MedDRA Version 16.0 terminology
Measure: Number; unit: participants
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 119 | 113
participants
  Total number of patients affected | 2 | 1
  Bradycardia and Hyperglycaemia | 1 | 0
  Haematemesis | 1 | 0
  Transient ischemic attack | 0 | 1

13. Other Pre Specified Outcome: Each Adverse Event (AE)
Description: Total number of patients affected.
Time Frame: Starting at Visit 2/ Start of Lead-In period (Day 7 up to day 119)
Population: 119 patients were randomized to Traumeel/Zeel and 113 patients to Placebo and all randomized patients were included in the Safety Set. 8 patients without any injection (not randomized) reported 12 adverse events
Measure: Number; unit: participants
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 119 | 113
participants | 64 | 43

14. Other Pre Specified Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs)
Description: Total number of patients affected.
Time Frame: during the treatment period and follow up period (Days 11 to 119)
Population: 119 patients were randomized to Traumeel/Zeel and 113 patients to Placebo and all randomized patients were included in the Safety Set. MedDRA Version 16.0 terminology. Adverse events during treatment (treatment-emergent) in 5% or more of total study patients
Measure: Number; unit: participants
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 119 | 113
participants
  Total Number of Patients affected | 64 | 43
  Musculoskeletal and connective tissue disorders | 26 | 14
  Infections and infestations | 12 | 10
  Nervous system disorders | 14 | 8
  Skin and subcutaneous tissue disorders | 14 | 9
  General disorders and administration site conditio | 11 | 8
  Injury, poisoning and procedural complications | 6 | 6

15. Other Pre Specified Outcome: Proportion of Patients Who Discontinued Due to an AE
Description: Total number of patients affected.
Time Frame: All visits (Days 1 up to 119)
Population: 119 patients were randomized to Traumeel/Zeel and 113 patients to Placebo and all randomized patients were included in the Safety Set. Medical Dictionary for Regulatory Activities (MedDRA) Version 16.0 terminology.
Measure: Number; unit: participants
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 119 | 113
participants
  Total number of patients affected | 3 | 4
  Injection site joint pain | 1 | 1
  Injection site vesicles | 1 | 0
  Haemarthrosis | 1 | 0
  Muscle tightness | 0 | 1
  Pain in extremity | 0 | 1
  Nephrolithiasis | 0 | 1
  Rash maculopapular | 0 | 1

16. Secondary Outcome: Time to 50% Pain Relief (Study Population Measure Statistically Derived)
Description: Changes of the target (treated) knee pain following a 50 feet walk self-assessed by the patients on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) where 0 corresponded to 'None' and 100 to 'Extreme'. The time to 50% pain relief were statistical exercises and were analyzed for each individual patient from their self-assessment.
Time Frame: Statistically derived
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
days
  After 1st Injection | 15 [15 to 22] | 22 [15 to 23]
  After 2nd Injection | 22 [15 to 35] | 34 [22 to 54]
  After 3rd Injection | 29 [22 to 37] | 50 [36 to 64]
Statistical Analysis 1: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; After first injection of study drug; Test type: Superiority or Other; p = 0.2164, Log Rank; Results of Kaplan-Meier Analysis with p-value from 2-sided log-rank test for equality of survival functions
Statistical Analysis 2: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; After second injection of study drug; Test type: Superiority or Other; p = 0.1651, Log Rank — Results of Kaplan-Meier Analysis with p-value from 2-sided log-rank test for equality of survival functions
Statistical Analysis 3: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; After third injection of study drug; Test type: Superiority or Other; p = 0.2220, Log Rank; Results of Kaplan-Meier Analysis with p-value from 2-sided log-rank test for equality of survival functions

17. Secondary Outcome: Patients Achieving 100% Pain Relief
Description: Changes of the target (treated) knee pain following a 50 feet walk self-assessed by the patients on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) where 0 corresponded to 'None' and 100 to 'Extreme'. The time to 100% pain relief were statistical exercises and were analyzed for each individual patient from their self-assessment, however, the prevalence of 100% pain relief did not support an estimate for the median time. The number of patients who reached 100% pain relief is reported and the log rank test for difference in time to 100% pain relief was calculated for each injection.
Time Frame: Statistically derived
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
participants
  After 1st Injection | 26 | 12
  After 2nd Injection | 25 | 12
  After 3rd Injection | 26 | 11
Statistical Analysis 1: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; After first injection of study drug; Test type: Superiority or Other; p = 0.0264, Log Rank; For equality of survival functions
Statistical Analysis 2: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; After second injection of study drug; Test type: Superiority or Other; p = 0.0346, Log Rank; For equality of survival functions
Statistical Analysis 3: Comparison: Co-administered Traumeel® and Zeel® vs Placebo Injectable Solution; After third injection of study drug; Test type: Superiority or Other; p = 0.0172, Log Rank; For equality of survival functions

18. Secondary Outcome: Time to and Use of Rescue Medication (Acetaminophen up to 3000 mg Per Day for Breakthrough Pain) (Study Population Measure Statistically Derived) - Patients Use
Description: Time to and use of rescue medication (acetaminophen up to 3000 mg per day for breakthrough pain) as reported by the patients. Patients who used any rescue medication during the study.
Time Frame: Statistically derived
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
participants | 82 | 72

19. Secondary Outcome: Time to and Use of Rescue Medication (Acetaminophen up to 3000 mg Per Day for Breakthrough Pain) (Study Population Measure Statistically Derived). Tablets Taken.
Description: Time to and use of rescue medication (acetaminophen up to 3000 mg per day for breakthrough pain) (study population measure statistically derived). Total number of tablets taken as reported by patient.
Time Frame: Statistically derived
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Tablets
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Number analyzed (Participants) | 117 | 111
Tablets | 49.0 (64.64) | 55.8 (59.71)

ADVERSE EVENTS:
Time Frame: Study Duration, 9 Months.
Description: The safety analysis included 232 randomized patients receiving at least one injection. 119 patients were randomized to Traumeel/Zeel and 113 patients to Placebo
Arm/Group | Co-administered Traumeel® and Zeel® | Placebo Injectable Solution
Serious Adverse Events (participants affected / at risk) | 2/119 | 1/113
Other Adverse Events (participants affected / at risk) | 64/119 | 43/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-administered Traumeel® and Zeel® (N=119) | Placebo Injectable Solution (N=113)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Co-administered Traumeel® and Zeel® (N=119) | Placebo Injectable Solution (N=113)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 8
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Joint crepitation (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gingival abscess (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pyoderma (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 10 | 3
Presyncope (Nervous system disorders) | 2 | 1
Sciatica (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 0 | 2
Burning sensation (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Injection site joint pain (General disorders) | 4 | 1
Pain (General disorders) | 5 | 0
Injection site vesicles (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 2
Injection site bruising (General disorders) | 1 | 0
Injection site erythema (General disorders) | 0 | 1
Injection site joint swelling (General disorders) | 0 | 1
Injection site scab (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Spinal pain (General disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Blood pressure increased (Investigations) | 1 | 1
Blood urine present (Investigations) | 0 | 1
Eosinophil count increased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Red blood cell count increased (Investigations) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Dacryostenosis acquired (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Lenticular opacities (Eye disorders) | 0 | 1
Presbyopia (Eye disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agreements in place restricting the PI from independently publishing the study results.